CLINICAL TRIAL: NCT02034266
Title: Phase 2 Study of the Effects of Omega-3 Fatty Acid Supplementation on Nerve Structure and Function in Type 1 Diabetes Mellitus - A Clinical Pilot Study
Brief Title: The Effect of Omega-3 Supplementation on Nerve Structure and Function in Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eduardo Ng (Other)
Collaborators: Canadian Diabetes Association (Other)
Responsible Party: Sponsor-Investigator, Eduardo Ng, Clinical Research Manager, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: T1DM Omega-3 study
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Type 1 Diabetes
Keywords: Type one diabetes; nerve damage; neuropathy; omega-3 fatty acid; supplementation; nutrition
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: open label study with no placebo.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omega-3 supplementation (Experimental): Participants will take an oral 5 mL serving (1 tbsp) of mammalian omega-3 seal oil (375 mg EPA, 280 mg DPA and 510 mg DHA) (Auum Inc., Timmons, On) twice daily. Total daily essential fatty acid load - 2330 mg.
  Interventions: Dietary Supplement: Omega-3 supplementation

INTERVENTIONS:
Dietary Supplement: Omega-3 supplementation — 5 mL twice daily, administered under the tongue
  Other Names: Auum Omega-3 oil

SUMMARY:
Nerves are made of different fats including omega-3s and omega-6s; however, dietary intakes of omega-6s are very high and omega-3 intakes are very low. We hypothesize that omega-3 supplementation will stop diabetes related changes in cornea nerve structure in patients with type 1 diabetes to stop the development of nerve injury associated with future risk of neuropathy, and reflect changes in the degree of nerve injury over time. As such, we anticipate that patients in the study will maintain Corneal Nerve Fiber Length (CNFL), the primary outcome measure.

DETAILED DESCRIPTION:
This study will test the use of an omega-3 supplement as a potential way to stop nerve damage that has been observed in individuals with type 1 diabetes Nerves supply signals to all structures in the body and take signals back to the spinal cord and brain. Both small and large nerve fibres can be affected in disease states, such as diabetes. Since defects of small nerve fibre activity have important consequences (painful symptoms, erectile dysfunction, cardiac rhythm disturbances, bladder and gastrointestinal dysfunction), it is important to determine new ways to maintain their function to help individuals maintain a high quality of life.

Until now, researchers have only tested the effect of omega-3 supplementation in animals with diabetes and have found this nutrient to lessen nerve damage while maintaining the function of nerves. However, there has not been any research on the use of omega-3s on nerve structure and function in humans with type 1 diabetes.

Current standard of care for type 1 diabetes is to manage glycemic control and any painful symptoms through medication. The use of omega-3 supplements for prevent or limit nerve damage in diabetes is not within the current standard of care. In this study omega-3 supplementation is experimental and has been approved by Health Canada for use in this study.

ELIGIBILITY:
Inclusion Criteria:

A. Patients of any gender or race aged 18 or above B. Type 1 diabetes mellitus as defined by the 2008 Canadian Diabetes Association C. Toronto Clinical Neuropathy Score ≥1 D. Ability to understand and cooperate with study procedures

Exclusion Criteria:

A. Current eye infection or damage of cornea B. Severe movement disorder C. History of allergy to proparacaine (the ocular topical anaesthetic used for the corneal confocal microscopy exam) D. Inability to sit and lie supine comfortably for 45-60 minutes E. Major medical or psychiatric illness that would preclude successful participation in the study F. Unwillingness to sign informed consent. G. Confirmed neuropathy secondary to non-diabetic causes (examples include polyneuropathy owing to alcohol abuse, B12 deficiency, folate deficiency, chronic renal failure, hypothyroidism, or neurotoxic drug use such as chemotherapy).

H. Current or previous regular (>3 times per week) consumption of omega-3 supplements within the past month I. Consistently consuming fish >2 times per week in the past month J. Performing regular exercise >3 times per week in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in corneal nerve fibre length | Baseline and 12 months
  Participants will undergo examination of nerve fibres adjacent to the Bowman's layer of the cornea in both eyes using the Rostock Cornea Module of the Heidelberg Tomograph III (Heidelberg Engineering, Smithfield RI, USA) to determine corneal IVCM corneal nerve fibre length (CNFL).

SECONDARY OUTCOMES:
Nerve Conduction Studies | Baseline and 12 months
  Nerve conduction studies will be conducted using standardized testing of the left median, ulnar, peroneal, and sural sensory nerves for signal amplitude and conduction velocity.
Corneal Nerve Fibre Length | 4 months and 8 months
  Interim measures of CNFL will be measured as a secondary outcome to track progressive changes with supplementation.
Laser Doppler Imaging Flare (LDI Flare) sympathetic skin response | Baseline and 12 months
  The purpose of this measure is to document, separate from the corneal IVCM parameters, small nerve fiber function. LDI Flare measurement will be conducted on MoorLDI2 Laser Doppler blood perfusion imager.
Vibration Perception Threshold | Baseline and 12 months
  Vibration perception threshold will be performed using the Neurothesiometer to evaluate sensory nerve function.
Cooling Detection Threshold Testing | Baseline and 12 months
  Cooling detection threshold testing will evaluate peripheral sensory nerve function.
Omega-3 status | Baseline, 4, 8 and 12 months
  Red blood cell omega-3 content will be determined using gas-flame chromatography.
Heart Rate Variability | Baseline and 12 months
R-R interval | Baseline and 12 months

OTHER OUTCOMES:
Glycated hemoglobin A1c | Baseline and 12 months
  Measure of glycemic control
Serum lipids | Baseline and 12 months
Thyroid stimulating hormone | Baseline and 12 months
Creatinine | Baseline and 12 months
Vitamin B12 | Baseline and 12 months
Serum Folate | Baseline and 12 months
Uric acid | Baseline and 12 months
Urinary albumin excretion | Baseline and 12 months
Serum protein electrophoresis | Baseline and 12 months
Serum C-reactive protein | Baseline and 12 months
Serum fatty acid profile | Baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vera Bril, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Division of Neurology, Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Lewis EJH, Perkins BA, Lovblom LE, Bazinet RP, Wolever TMS, Bril V. Effect of omega-3 supplementation on neuropathy in type 1 diabetes: A 12-month pilot trial. Neurology. 2017 Jun 13;88(24):2294-2301. doi: 10.1212/WNL.0000000000004033. Epub 2017 May 17. PMID 28515269